CLINICAL TRIAL: NCT06100029
Title: The Effect of Lavender Essential Oil for Delirium in Elderly Intensive Care Unit Patients: Study Protocol for a Double Blind, Randomized, Placebo-controlled Trial
Brief Title: The Effect of Lavender Essential Oil for Delirium in Elderly Intensive Care Unit Patients: Study Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Traditional Chinese Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ChongqingTCMH
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Delirium in Old Age
MeSH Terms: interventions — lavender oil; Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): lavender aromatherapy
  Interventions: Drug: Lavender; Behavioral: A2F bundle
- Control group (Placebo Comparator): distilled water
  Interventions: Behavioral: A2F bundle

INTERVENTIONS:
Drug: Lavender — The lavender aroma (L. angustifolia ssp. Angustifolia) is provided by Pranarom International, Ghislenghien, Belgium. Lavender aroma will be contained in a 10 ml glass bottle with a drop stopper and place the bottle within 20 cm of the patient's pillow so that the aroma can reach the patient. The entire course of treatment lasts 5 days.
  Other Names: aromatherapy
  Arms: Intervention group
Behavioral: A2F bundle — A: assess, prevent, and manage pain; B: both spontaneous awakening and breathing trials; C: choice of analgesia and sedation; D: delirium assessment, prevention, and management; E: early mobility and exercise; and F: family engagement/empowerment
  Other Names: ABCDEF bundle

SUMMARY:
Elderly critically ill patients in the intensive care unit (ICU) are at risk of delirium, which is primarily characterized by acute consciousness impairment and perceptual, cognitive, and memory impairment, resulting in excess death, care expenditures, and acquired dementia, depression and anxiety, which severely affect the prognosis of critically ill patients. However, there are currently no effective pharmacological strategies for preventing delirium. Inhalation aromatherapy has been proven to benefits the sleep disorder, anxiety or depression and lavender oil is one of the most used essential oils. Therefore, we hypothesized that the use of lavender would reduce the incidence rate of delirium in ICU patients.

DETAILED DESCRIPTION:
This trial was designed to be a randomized, single-center, double-blind, placebo-controlled trial. A total of 68 elderly patients from two ICUs will be randomly allocated at a 1:1 ratio to the intervention group or the control group. Both groups will receive the ABCDEF (A2F) bundle strategy recommended by guidelines, a multicomponent approach including pain and delirium management, breathing trial practice, analgesic and sedation usage control, family engagement and so on, to prevent delirium. The intervention group will additionally receive aromatherapy lasting for five days. The primary outcome is the prevalence of delirium. Secondary outcomes include the severity and duration of delirium, the length of ICU stay, the duration of physical restraint, the duration of analgesic and sedative medication and the 28-day mortality rate. We will use the CAM-ICU and CAM-S to measure the prevalence and severity of delirium, and analyses of variance (ANOVAs) or repeated-measures ANOVAs and Wilcoxon rank-sum tests to analyze the observation results.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients aged between 60 and 90 years old
* Had an expected total ICU length of stay (LOS) of 72 hours or more
* Admitted to the ICU within 48 hours before screening
* Signed the informed consent form.

Exclusion Criteria:

* Incapacitation preventing the assessment of delirium (i.e., coma, sedation, or active seizures)
* History of psychiatric disorders, dementia, Parkinson's disease, use of antipsychotic drugs, or alcohol dependence
* History of traumatic brain injury or brain infection
* Diagnosis of delirium prior to intervention initiation
* Allergies to medications used in the protocol or current participation in other drug studies
* Inability to communicate in Chinese or English
* Expected to be discharged or deceased within 72 hours of admission.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
the prevalence of delirium | Through study completion, an average of 1 year (November 31, 2023-November 31, 2024)
  Assessment will be performed during the study period for all enrolled participants in a timely manner using the Confusion Assessment Method for the ICU (CAM-ICU). The CAM-ICU, a 2-minute assessment tool, has proven to be quick, valid, and reliable for the diagnosis of delirium in the ICU, making it beneficial for use in both clinical and research contexts.

SECONDARY OUTCOMES:
Severity of delirium | Through study completion, an average of 1 year (November 31, 2023-November 31, 2024)
  Throughout the study, the Confusion Assessment Method-Severity scale will be administered in each included patient. The total score of the Confusion Assessment Method-Severity scale can vary between 0 and 7, where 7 indicates the most severe condition.
Duration of delirium | Through study completion, an average of 1 year (November 31, 2023-November 31, 2024).
  Once delirium is diagnosed, the investigators will record its duration of the patient tests positive for the Confusion Assessment Method for the ICU (CAM-ICU)

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Ren, Study Director — Chongqing Traditional Chinese Medicine Hospital
Locations (1):
- Chongqing traditional Chinese medicine hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: No